CLINICAL TRIAL: NCT02875951
Title: Prospective, Non-interventional, Non-controlled Multicenter Observational Study to Evaluate Aspects of Pharmaceutical Care and the Treatment of Postmenopausal Patients With Hormone-receptor Positive, HER2-receptor Negative, Advanced Breast Cancer Treated With Everolimus and Exemestane.
Brief Title: Investigating Patient Satisfaction With Oral Anti-cancer Treatment in Patients With Hormone-receptor Positive, HER2-receptor Negative, Advanced Breast Cancer
Acronym: IPSOC-mamma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Sandra De Coster, Pharmacist, KU Leuven
Other Study IDs: VF/2014/03
Record Dates: First submitted 2016-07-18; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: ER Positive, HER2 Negative Breast Cancer Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ER positive, HER2 negative breast cancer patients: Postmenopausal patients with hormone receptor positive, HER2 receptor negative breast cancer

SUMMARY:
A prospective, non-interventional, non-controlled multicenter observational study to evaluate aspects of pharmaceutical care and the treatment of postmenopausal patients with hormone-receptor positive, HER2-receptor negative, advanced breast cancer treated with everolimus and exemestane.

The main objective of the study is to evaluate medication adherence in postmenopausal, hormone-receptor positive, HER2-receptor negative, advanced breast cancer treated with a combination of everolimus and exemestane. Additionally, other aspects of the pharmacotherapy, with focus on the patient perspective, will be investigated:

* Patient satisfaction with treatment information
* Patient satisfaction with treatment
* Health-related quality of life
* Treatment efficacy
* Treatment-related toxicity
* Patient follow-up by the oncologic team/general practitioner and or specialized home nurses

This study should reveal information necessary for the development of pharmacotherapeutic care concepts that meet the needs of cancer patients treated with an oral anti-cancer drug over a long period.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, 18 years or older
* Signed written informed consent
* Patient can be contacted by phone and/or e-mail
* HR+, HER2- advanced or metastatic breast cancer
* Recurrence or progression following a non-steroidal aromatase inhibitor
* Able to swallow and retain oral medication
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2

Exclusion Criteria:

* Patients who are not able to understand Dutch or French
* Symptomatic visceral metastatic disease
* Patients who have taken an investigational drug within 28 days or 5 half-lives, whichever is shorter, prior to recruitment
* Current use of a prohibited medication as described in the SPC
* Any serious or unstable pre-existing medical conditions, psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedure
* Hypersensitivity to the active substances or to any of the excipients

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postmenopausal women with hormone-receptor positive, HER2 receptor negative advanced breast cancer, without symptomatic visceral disease after recurrence or progression following a non-steroidal aromatase inhibitor, starting with a combination treatment of everolimus & exemestane
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | one year
  At the first visit patients will receive their anti-cancer medication by the hospital in two separate pill boxes which electronically record openings cf. Medication Event Monitoring System (MEMS®, Aardex). The recorded information in these chips will be read in the hospital pharmacy each time the patient gets new capsules. This information is strictly confidential and can only be consulted by the research team at the KULeuven.

SECONDARY OUTCOMES:
Patient Satisfaction with Cancer Treatment Education (Ps-CaTE) | one year
  Satisfaction with cancer treatment information will be assessed, using a standardised questionnaire at the start of the treatment and after approximately 1, 3, 6 and 12 months of treatment
Morisky Medication Adherence Scale (MMAS) | one year
  Medication adherence will be assessed, using a standardised questionnaire, after approximately 1, 3, 6 and 12 months of treatment.
Cancer Therapy Satisfaction Questionnaire (CTSQ) | one year
  Satisfaction with cancer treatment will be assessed, using a standardised questionnaire, after approximately 1, 3, 6 and 12 months of treatment.
Functional Assessment of Cancer Therapy - for patients with breast cancer (FACT-B) | one year
  Health-related quality of life will be assessed, using a standardised questionnaire, at the start of the treatment and after approximately 1, 3, 6 and 12 months of treatment.
Tumor status evaluation | one year
  Tumor status evaluation of the patient will be assessed by the treating oncologist by CA15-3 & CEA markers at the start of the study and after 1, 3, 6 and 12 months of treatment.
Tumor status evaluation | one year
  Tumor status evaluation of the patient will be assessed by the treating oncologist by RECIST criteria after 1, 3, 6 and 12 months of treatment.
Performance status of the patient | one year
  Performance status of the patient will be assessed by the treating oncologist by ECOG criteria at the start of the study and after 1, 3, 6 and 12 months of treatment.
Toxicity of treatment | one year
  Severity of adverse events and relation to the treatment will be assessed by the treating oncologist, based on CTC-NCI 4.0, after 1, 3, 6 and 12 months of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Katholieke Universiteit Leuven - Clinical Pharmacology and Pharmacotherapeutics, Leuven, Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No